CLINICAL TRIAL: NCT03746470
Title: A Randomized Controlled Trial to Evaluate the Graft Ligamentization and Integration in the Reconstruction of the Anterior Cruciate Ligament With or Without Detachment of Hamstring Tendon Tibial Insertion
Brief Title: A Study to Compare Two Techniques for the Reconstruction of the Anterior Cruciate Ligament
Acronym: ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-003
Record Dates: First submitted 2018-10-30; First posted 2018-11-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Complete Tear, Knee, Anterior Cruciate Ligament
Keywords: arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insertion preserving (Experimental): ACL reconstruction preserving insertion
  Interventions: Procedure: ACL reconstruction preserving insertion
- insertion detaching (Active Comparator): ACL reconstruction detaching insertion
  Interventions: Procedure: ACL reconstruction detaching insertion

INTERVENTIONS:
Procedure: ACL reconstruction preserving insertion — Anterior cruciate ligament reconstruction with semitendinosus and gracilis, preserving their insertion at the level of the hamstring.
  Arms: insertion preserving
Procedure: ACL reconstruction detaching insertion — Anterior cruciate ligament reconstruction with semitendinosus and gracilis tendons completely detached from their insertion at the hamstring.
  Arms: insertion detaching

SUMMARY:
This is a prospective and randomized trial to compare two different techniques used in normal practice for the reconstruction of the anterior cruciate ligament in arthroscopy.

The experimental group (group 1) will undergo a reconstruction technique where semitendinosus and gracilis will preserve their insertion at the level of the hamstring whereas in the control group (group 2) the semitendinosus and gracilis tendons will be disengaged from their insertion on the hamstring .

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55
* MRI confirmed primary and total ACL injury of traumatic origin
* Indication for ACL reconstruction in arthroscopy
* Written informed consent
* Active and non-sedentary lifestyle

Exclusion Criteria:

* Complex meniscal injuries
* Cartilage lesions of sizes> 2 cm2
* Other ligamentous lesions
* Axis deviations greater than 10°
* Rheumatic, neuromuscular or general systemic diseases
* Prevention of injured knee traumas treated surgically
* Difficulties in compliance in following the rehabilitation programs
* Obesity (BMI ≥ 30)
* Neoplastic diseases, metabolic diseases, inflammatory and systemic diseases, autoimmune diseases, immunocompromised patients

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Graft integration by the Signal / Noise Quotient (SNQ) at 6 months | 6 months after ACL reconstruction intervention
  Signal intensity of the graft evaluated by the Signal / Noise Quotient (SNQ) during MRI 3 Tesla

SECONDARY OUTCOMES:
Graft integration by the Signal / Noise Quotient (SNQ) at 3 and 12 months | 3, 12 months after ACL reconstruction intervention
  Signal intensity of the graft evaluated by the Signal / Noise Quotient (SNQ) during MRI 3 Tesla
Right anatomical graft position | 12 months after ACL reconstruction intervention
  Evaluation of right anatomical graft position by MRI 3 TESLA
Anterior tibial translation | 3, 6, 12 months after ACL reconstruction intervention
  Anterior tibial translation will be measured in millimeters using the arthrometer Rolimeter
Anterior knee joint instability | 3, 6, 12 months after ACL reconstruction intervention
  Anterior knee joint instability will be measured by the device KiRA (Kinematic Rapid Assessment) by the parameters of the pivot-shift test
IKDC (International Knee Documentation Committee) questionnaire | 3, 6, 12 months after ACL reconstruction intervention
  Test to evaluate post-surgery instability with a scores range from 0 points to 100 points; patients report symptoms, sports and daily living activities
Tegner activity scale | 3, 6, 12 months after ACL reconstruction intervention
  Test to evaluate post-surgery instability with a scores range from 0 points to 10 points; patients describe their current level of activity and that before injury.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Decogliano, MD, Study Chair — EOC - Unità Traumatologia e Ortopedia - ORL
Locations (2):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy
- EOC - Unità Traumatologia e Ortopedia ORL, Lugano, Switzerland